CLINICAL TRIAL: NCT03422562
Title: Do Probiotics Modulate the Intestinal Microbiome of Extremely Preterm Infants?
Brief Title: Probiotics and Intestinal Microbiome in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Belal Alshaikh (Other)
Responsible Party: Sponsor-Investigator, Belal Alshaikh, Neonatologist, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: REB16-0542
Record Dates: First submitted 2018-01-10; First posted 2018-02-05 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-04

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Florababy probiotic (0.5g per day) will be started at or after 72 hours of life and will be administered in 1ml sterile water prior to feed.
  Interventions: Dietary Supplement: Florababy
- Control (No Intervention): Standard of care arm

INTERVENTIONS:
Dietary Supplement: Florababy — Probiotic supplement
  Arms: Probiotic

SUMMARY:
The gut microbiome plays a significant role in balancing the inflammatory system in the immature gut. A breakdown in this balance with altered colonization of the microbiota in very low birth weight (VLBW) preterm infants is associated with increased feeding intolerance, necrotizing enterocolitis (NEC) and sepsis. Probiotics are proposed to normalize microbial populations and decrease intestinal disease in preterm infants. There is limited data linking clinical outcomes with the biology of probiotics. We aim to study the colonization of the GI tract with probiotic species contained in a specific probiotic blend - Florababy - in VLBW preterm infants.

Stool microbiome will be analyzed at 4 time points in 2 groups (one given Florababy and the other no) of infants less than 1000 grams birth weight and < 29 weeks gestation. A comparison of stool microbiome analysis and the incidence of feeding intolerance and time to reach full feeds in the two groups will be made.

ELIGIBILITY:
Inclusion Criteria:

* Infants born less than 29 weeks gestation and <1000 g birth weight admitted to the Neonatal Intensive Care Unit (NICU) at Foothills Medical Centre in Calgary.

Exclusion Criteria:

* Infants with major congenital anomalies, hypoxic-ischemic injury, NEC or bowel perforation before 72 hours of life.

Ages: 23 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Stool Microbiome | 4 weeks
  difference in stool microbiome after Florababy or no drug administration

SECONDARY OUTCOMES:
Stool Microbiome | 2 weeks
  difference in stool microbiome after Florababy or no drug administration
Feeding intolerance | 4-6 weeks
  Incidence of feeding intolerance
Full Feeds | 4-6 weeks
  Time to reach full feeds.

CONTACTS AND LOCATIONS:
Overall Officials: Belal Alshaikh, MD, Principal Investigator — University of Calgary; Belal Alshaikh, MD, Principal Investigator — Physician
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alshaikh B, Samara J, Moossavi S, Ferdous T, Soraisham A, Dersch-Mills D, Arrieta MC, Amin H. Multi-strain probiotics for extremely preterm infants: a randomized controlled trial. Pediatr Res. 2022 Dec;92(6):1663-1670. doi: 10.1038/s41390-022-02004-z. Epub 2022 Mar 21. PMID 35314794

DOCUMENTS (3):
  • Study Protocol (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03422562/Prot_001.pdf
  • Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03422562/SAP_002.pdf
  • Informed Consent Form (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT03422562/ICF_000.pdf